CLINICAL TRIAL: NCT05938972
Title: Real Life Study Assessing Long Term Outcomes and Predictive Factors of Response to Biologicals in Patients With Severe CRSwNP and/or Severe Allergic and/or Eosinophilic Asthma
Brief Title: Real Life Study of Biologicals in Patients With Severe CRSwNP
Acronym: NASUMAB
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2022-0033
Record Dates: First submitted 2023-06-13; First posted 2023-07-11 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
MeSH Terms: interventions — mepolizumab; Omalizumab; dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — blood samples, nasal secretions and small tissue biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Mepolizumab — Monoclonal antibodies
  Other Names: Omalizumab; Dupilumab

SUMMARY:
This study is a pragmatic, real-life, observational study recruiting adult patients with chronic rhinosinusitis with nasal polyposis who are eligible to start biologicals as standard treatment. The aim of this study is to observe the long-term outcomes of biologicals in CRSwNP patients with or without comorbid asthma in 'real life'. Moreover, the investigators will gain insight into the mechanisms of biologicals in the local and systemic immunity of these patients and investigate novel local and systemic biomarkers and predictors of response.

DETAILED DESCRIPTION:
In this project, thanks to intense collaboration between the ENT department and the pulmonary diseases within the Allergy Network UZ Gent, the investigators set up a prospective study and biobank with the following aims:

* To observe and follow-up on clinical characteristics in patients with chronic rhinosinusitis with nasal polyposis (CRSwNP) with or without asthma. Primary outcomes will be the endoscopic total nasal polyp score (NPS) and the nasal symptom scores (SNOT-22, VAS, NCS and UPSIT).
* Identifying key nasal inflammatory biomarkers to predict therapeutic response to biologicals in CRSwNP patients (identification on blood samples, nasal secretions, small tissue biopsies and superficial scrapings before, during and at month 24 of treatment).
* Unravel the effects of biologicals in the local nasal immune regulation.
* Performing additional analyses to search for new biomarkers via complete proteomic analysis.

Using a unique combination of nasal sampling and state of the art biomarker discovery, the investigators believe this research will provide unprecedented insights which will aid the treatment of patients with biologicals.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria to be eligible for the enrolment in the study:

* Signed informed consent form (ICF),
* Age between 18 and 80 years at time of signing ICF,
* Able to comply with the study protocol, in the investigator's judgment,
* In group one: patients with severe allergic and/or eosinophilic asthma, defined by being currently treated with a biological (SoC) OR starting treatment with a biological (SoC).
* In group two: patients with CRSwNP with or without asthma, defined by starting treatment with a biological (SoC) and fulfill the criteria for reimbursement of a biological therapy

Exclusion Criteria:

Patients who do not meet the reimbursement criteria of a biological therapy cannot participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (between 18 and 80 years old) with severe allergic and/or eosinophilic asthma in group 1 and CRSwNP in group 2 that are receiving or will start to receive a biological as standard of care treatment, and agree on participating (signature of a written informed consent).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical characteristics | 24 months
  Endoscopic total nasal polyp score to quantify nasal polyps with endoscopy. The higher the score, the more polyps are present in the nose. A unilateral score from 0 (absence of polyps) to 4 is given. The total nasal polyp score is the sum of the scores for both nostrils, thus ranging from 0 to 8, and is based on the continuous extension of nasal polyps beyond clear landmarks such as the upper and lower borders of the middle and inferior turbinate. This implies that a score can only be attributed if the criteria of the lower scores are met. E.g. a unilateral score of 3 cannot be given without nasal polyps also meeting the criteria for a score of 2, and similarly, a score of 4 cannot be given without having a score of 3.
Clinical characeristics | 24 months
  Nasal symptom scores: VAS symptom scores and SNOT-22 questionnaire will be recorded through a questionnaire. The need for surgery or rescue medication (e.g. Systemic corticosteroids, antibiotics,..) will be recorded each study visit.
  1. VAS symptom score: minimum of 0 to maximum of 100. Higher VAS-scores indicate worse symptoms.
  2. SNOT-22 score: a validated, self-administered questionnaire that is used to assess CRS patients. It consists of 22 items, rated from 0 ('no problem at all') to 5 ('worst possible symptom'). Possible SNOT-22 total scores range from 0 to 110, with higher SNOT-22 total scores indicating worse symptoms
Local nasal immunity | 24 months
  Nasal secretions will be harvested at each visit. Merocels (IVALON 4000 Plus 3,5 x 0,9 x 1,2 cm surgical products Fabco, New London, CT) will be placed in each nostril for 5 minutes and will be stored at -20°C until analysis. Key inflammatory markers will be measured: ECP, IL-5, sIL-5Rα, total IgE, periostin, total lambda- and kappa-FLC concentrations, MMP-9 and MPO. Additional analyses will then be performed to search for new biomarkers via complete proteomic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gevaert, Prof. Dr., Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided